CLINICAL TRIAL: NCT01411839
Title: Addressing Depression and ART Adherence in HIV+ Latinos on the U.S.-Mexico Border
Brief Title: Depression and ART Adherence in HIV+ Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Texas (Other)
Responsible Party: Principal Investigator, Jane Simoni, Professor, Psychology; Adjunct Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35279; R34MH084674 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-08-08 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Depressive Symptoms; HIV Infections
Keywords: Depression; Latinos; Adherence; Cognitive-Behavioral Therapy; HIV/AIDS
MeSH Terms: conditions — Depression; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-Behavioral Therapy (CBT-AD) (Experimental): This arm type is a cognitive-behavioral therapy program intervention for issues of medication adherence and depression. The intervention is a therapy program intervention involves 10-weekly or biweekly sessions, with 2 booster session, and focused on psychoeducation, behavioral activation, cognitive restructuring, and problem-solving. A letter was sent to their medical provider indicating that mild symptoms of depression were detected and that they were enrolled in this intervention, but no details were provided regarding their assignment to one of two conditions/arms.
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT-AD)
- Control-Standard Care (No Intervention): Those randomized to the control condition are not involved in the CBT-AD therapy intervention. They receive standard care as usual. A letter was sent to their medical provider indicating that mild symptoms of depression were detected and that they were enrolled in this intervention, but no details were provided regarding their assignment to one of two conditions/arms. The participants in the control arm are followed and matched to a participant in the intervention arm.

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT-AD) — CBT-AD is a therapy program intervention that uses one-on-one and face-to-face patient-therapist sessions.
  Other Names: CBT-AD
  Arms: Cognitive-Behavioral Therapy (CBT-AD)

SUMMARY:
The current HIV treatment adherence project was designed to adapt culturally and then pilot test an empirically supported cognitive-behavioral therapy program for adherence and symptoms of depression (CBT-AD)with HIV+ Latinos living on the U.S.-Mexico Border.

DETAILED DESCRIPTION:
Additionally, the investigators will assess the feasibility and efficacy of a novel medication monitoring and reminder system (MedSignals®) in the form of an electronic pillbox with monitoring and reminding functions that is available in a Spanish-language version. Our hypotheses are grounded in a conceptual model proposing that the CBT-AD intervention will improve problem-solving ability and decrease depressive symptomatology, which will directly improve biomedical outcomes of HIV-1 RNA viral load and CD4 as well as indirectly improve biomedical outcomes through increased motivation, improved memory, and better medication adherence. Evaluating and implementing generalizable and sustainable mental health and adherence interventions such as the ones proposed are urgently needed in the region to improve HIV treatment outcomes and thwart the development and transmission of drug resistant virus.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ participants (a) currently receiving HIV care at La Fe CARE Center (study site);
* 18 years of age or older;
* Latino (i.e., self-identified as being of Mexican heritage);
* English- or Spanish-speaking
* capable of giving informed consent;
* currently on a prescribed antiretroviral regimen;
* suboptimally adherent (i.e., demonstrated either by a VL load taken in the last 12 months that is above the undetectable threshold of 50 mL copies or self-reporting a missed dose in the last two weeks);
* exhibiting some depressive symptomatology (i.e., scoring on the Beck Depression Inventory-1A 10 or above), and (i) male or female (including transgender Female-to-Male and Male-To-Female.

Exclusion Criteria:

* actively psychotic or so cognitively impaired that they cannot participate,
* so physically ill as to be unable to come to the clinic to participate in the intervention, OR
* Report The use of crack, cocaine, heroin, OR methamphetamines to any extent in the past 40 days.
* Those who are planning on being away from the area for any extended period during the study (as in the case of seasonal workers) or whom
* have household members already enrolled in the study will also be excluded. We did choose to restrict study eligibility to individuals of Mexican descent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane M Simoni, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Centro de Salud Familiar La Fe CARE Center, El Paso, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected in a two-stage process from 10/21/2009 - 8/31/2011 at a publicly-funded community health clinic in El Paso, TX, on the U.S.-Mexico border.
Pre-assignment Details: Eligible participants were randomly assigned to the intervention or treatment as usual (TAU) control condition, both enhanced with the notification letter to provider. An external statistician had used a computerized random number generator to select random permuted blocks of four.
Groups:
- Cognitive-Behavioral Therapy (CBT-AD): CBT intervention for adherence and depression in a sample of HIV+ Latinos. The intervention is designed for issues of non-adherence and depressive symptomatology. Therapy intervention involves 10-weekly or biweekly sessions, with 2 booster session.
  Cognitive-Behavioral Therapy AD: Therapeutic intervention, one-on-one and face-to-fact, over multiple sessions
- Control-Standard Care: Those randomized to the control condition are not involved in the CBT-AD therapy intervention. They receive standard care as usual. A letter is sent to their medical provider indicating that mild symptoms of depression were detected. The participants in the control arm are followed and matched to a participant in the intervention arm.
Period: Overall Study
Arm/Group | Cognitive-Behavioral Therapy (CBT-AD) | Control-Standard Care
Started | 20 | 20
Completed | 16 | 17
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Therapy (CBT-AD) | Control-Standard Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (10.7) | 44.8 (10.7) | 46 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 20 | 40
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Beck Depression Inventory 1a [Mean (Standard Deviation); unit: units on a scale] — Self-reported depressive symptoms were assessed at each time point using the revised Beck Depression Inventory-Ia (BDI-Ia), which consists of 21 items, each with a 4-point response scale anchored with descriptive statements. Scores can range from 0-63, and scores of 10 or higher are presumptive of mild depressive severity. The BDI scores presented were added up and higher scores indicate worse depression.
  units on a scale | 22 (9.2) | 16.8 (6.3) | 19.4 (8.2)
Visual Analog Scale 30-day Adherence [Mean (Standard Deviation); unit: Percent of doses taken] — Self-reported adherence was assessed with the visual analog scale. This is a 10cm line that is shown to patients who then mark on the line (from 0 to 100% in 1cm intervals) how much medication they have taken. Higher scores indicate better adherence.
  Percent of doses taken | 84.4 (24.4) | 90.6 (11.1) | 87.2 (19.5)
Electronic Drug Adherence Monitoring [Mean (Standard Deviation); unit: Percent Adherence] — The MedSignals electronic pill-box is a storage bin that allows participants to store medications. In the treatment condition, the pill-box provides audio commands to alarm participants that it is time to take their medication. The pill-box stores adherence data (time, number of openings). In the control condition, the pill-box does not alarm participants but serves in the same capacity otherwise. All data is uploaded electronically. Higher numbers indicate better adherence that correspond to pill-box openings corresponding the designated time of taking their medication.
  Percent Adherence | 43.2 (43.5) | 55.6 (47.6) | 49.4 (40.6)
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a 10-item clinician administered scripted rating scale of depressive symptoms (each of the ten items is scored from 0-6, with total scores ranging from 0 to 60). The scale was developed to capture current depressive symptoms within the past seven days. The areas covered include: apparent and reported sadness, inner tension, reduced sleep and appetite, concentration difficulties, lassitude, inability to feel, pessimistic and suicidal thoughts. Higher scores indicate the presence of more depressive symptoms.
  units on a scale | 25.1 (9.7) | 22.1 (9.8) | 23.6 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Depression From (1) Clinician-Administered MADRS Measure, and (2) Participant Self-Report Ratings With BDI-1a
Description: 1. Clinician-administered ratings are scored on the MADRS. The MADRS is a 10-item, past 7-day clinician administered scripted rating scale of depressive symptoms (each of the ten items is scored from 0-6, with total scores ranging from 0 to 60). The areas are: apparent and reported sadness, inner tension, reduced sleep/appetite, concentration difficulties, lassitude, inability to feel, pessimistic and suicidal thoughts. Higher scores indicate the presence of more depressive symptoms.
  2. Participant self-report ratings are scored on the BDI-1a. The BDI-1a is assessed at each time point using the revised Beck Depression Inventory-Ia (BDI-Ia), which consists of 21 items, each with a 4-point response scale anchored with descriptive statements. Scores can range from 0-63, and scores of 10 or higher are presumptive of mild depressive severity. The BDI scores presented were added up and higher scores indicate worse depression. The MADRS and BDI-Ia is scored a total units on the scale.
Time Frame: MADRS and BDI-1a scores at 6 and 9-month follow-up
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cognitive-Behavioral Therapy (CBT-AD) | Control-Standard Care
Number analyzed (Participants) | 20 | 20
Units on a scale
  MADRS at 6-month follow-up | 17.8 (12.2) | 19.2 (11.2)
  MADRS at 9-month follow-up | 19.7 (12.7) | 17.7 (12.9)
  BDI-1a at 6-month follow-up | 15.0 (7.4) | 11.8 (7.0)
  BDI-1a at 9-month follow-up | 14.2 (7.0) | 13.5 (9.0)

2. Secondary Outcome: Self-Report Adherence
Description: Self-reported adherence was assessed with the visual analog scale (VAS). The VAS is a 10cm line that is shown to patients who then mark on the line (from 0 to 100% in 1cm intervals) how much medication they have taken. Higher scores indicate better adherence.
Time Frame: Self-reported adherence at 6 and 9-month follow-up
Measure: Mean (Standard Deviation); unit: Percent of all doses of medication taken
Arm/Group | Cognitive-Behavioral Therapy (CBT-AD) | Control-Standard Care
Number analyzed (Participants) | 20 | 20
Percent of all doses of medication taken
  Self-report adherence at 6-month follow-up | 92.6 (9.4) | 86 (14.7)
  Self-report adherence at 9-month follow-up | 93.5 (9.0) | 91.9 (7.7)

3. Secondary Outcome: MedSignals Electronic Pill-box for Adherence
Description: The MedSignals electronic pill-box is a storage bin that allows participants to store medications. In the treatment condition, the pill-box provides audio commands to alarm participants that it is time to take their medication. The pill-box stores adherence data (time, number of openings). In the control condition, the pill-box does not alarm participants but serves in the same capacity otherwise. All data is uploaded electronically. Higher numbers indicate better adherence that correspond to pill-box openings corresponding to the designated time of taking their medication.
Time Frame: 6 and 9 month follow-up adherence scores
Measure: Mean (Standard Deviation); unit: Percent adherence
Arm/Group | Cognitive-Behavioral Therapy (CBT-AD) | Control-Standard Care
Number analyzed (Participants) | 20 | 20
Percent adherence
  Electronic Adherence at 6-month Follow-Up | 45.8 (47.8) | 28.8 (31)
  Electronic Adherence at 9-month Follow-Up | 31.1 (44.9) | 20.0 (31.5)

ADVERSE EVENTS:
Time Frame: 1 Year, 9 Months.
Arm/Group | Cognitive-Behavioral Therapy (CBT-AD) | Control-Standard Care
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No